CLINICAL TRIAL: NCT00678886
Title: Durable-Response Therapy Evaluation For Early or New-Onset Type 1 Diabetes - DEFEND
Brief Title: Trial of Otelixizumab for Adults With Newly Diagnosed Type 1 Diabetes Mellitus (Autoimmune): DEFEND-1
Acronym: DEFEND-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115495; TRX4006 (Other: Tolerx); NCT00893022 (obsolete NCT alias)
Record Dates: First submitted 2008-05-13; First posted 2008-05-16 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; new onset type 1 diabetes; T1DM; Type l diabetes; juvenile diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antibodies, Monoclonal; otelixizumab; Muromonab-CD3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- otelixizumab (Experimental): otelixizumab
  Interventions: Biological: otelixizumab infusion plus physician determined standard of care
- placebo (Placebo Comparator): Placebo
  Interventions: Biological: placebo infusion plus physician determined standard of care

INTERVENTIONS:
Biological: otelixizumab infusion plus physician determined standard of care — infusion
  Other Names: monoclonal antibody; ChAglyCD3; anti-CD3; TRX4
  Arms: otelixizumab
Biological: placebo infusion plus physician determined standard of care — infusion
  Arms: placebo

SUMMARY:
The purpose of this study is to find out if an 8-day series of otelixizumab infusions leads to greater improvement in insulin secretion as compared with placebo infusion. Insulin secretion will be assessed using mixed meal-stimulated C-peptide.

Subjects will be assigned to receive either otelixizumab or placebo at a ratio of 2:1 (2/3 otelixizumab, 1/3 placebo). These study agents will be administered as an addition to insulin, diet, and other physician determined standard of care treatments.

DEFEND-1 is now closed to enrollment.

DEFEND-2 will begin early in 2010. It is very similar to DEFEND-1 and will again require subjects with new onset type 1 diabetes. Please check back here for more details.

In the meantime, established and new onset type 1 diabetes patients in North America are welcome to consider the TTEDD study:

http://www.clinicaltrials.gov/ct2/show/NCT00451321?term=TTEDD&rank=1

DETAILED DESCRIPTION:
The following visits are required:

* Screening Visits: 2 to 3 appointments will be conducted to determine eligibility. At 2 of these visits participants will drink a liquid meal and have blood tests done over the post-meal period.
* Dosing Visits: 8 outpatient visits on consecutive days, each lasting about 4-6 hours.
* Follow-up Visits: weekly for the first month, then every 2 weeks for 3 months, followed by monthly visits through 1 year. There will be 3 visits in the second year.
* The total duration of the study is 2 years.
* Glucose test strips, glucose monitors and PDAs to record insulin will be provided to all study subjects for the duration fo the study. Frequent glycemic monitoring will occur through lab testing and blood glucose self-monitoring to help facilitate tight glycemic control in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-45
* Diagnosis of diabetes mellitus, consistent with ADA criteria
* No more than 90 days between diagnosis and administration of study compounds
* Requires insulin for type 1 diabetes mellitus, or has required insulin at some time between diagnosis and administration of study compounds.
* Stimulated C-peptide level greater than 0.20 nmol/L and less than or equal to 3.50 nmol/L
* Positive for one or more of the autoantibodies typically associated with T1DM: antibody to glutamic acid decarboxylase (anti-GAD); antibody to protein tyrosine phosphatase-like protein (anti-IA-2); zinc transporter autoantibodies (ZNT8); insulin autoantibodies (IAA). A subject who is positive for insulin autoantibodies (IAA) and negative for the other autoantibodies will only be eligible if the subject has used insulin for less than 7 days total.

Exclusion Criteria:

* Other, significant medical conditions based on the study doctor's evaluation

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 272 (Actual)
Dates: Start 2008-07-29 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2012-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (101):
- United States (61):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Costa Mesa, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Trinity, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Atlanta, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Mentor, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Langhorne, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hurst, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Tacoma, Washington
- Canada (6):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Smiths Falls, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
- GSK Investigational Site, Arhus C, Denmark
- Finland (2):
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Germany (4):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Bad Nauheim, Hesse
  - GSK Investigational Site, Bad Lauterberg im Harz, Lower Saxony
  - GSK Investigational Site, Berlin
- Italy (6):
  - GSK Investigational Site, Latina, Lazio
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Monserrato, Sardinia
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Roma
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Sant Joan
  - GSK Investigational Site, Tarrasa, Barcelona
- Sweden (10):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Halmstad
  - GSK Investigational Site, Härnösand
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Karlstad
  - GSK Investigational Site, Kristianstad
  - GSK Investigational Site, Motala
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Vaxjo
- United Kingdom (6):
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Blackburn
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Background] Keymeulen B, Vandemeulebroucke E, Ziegler AG, Mathieu C, Kaufman L, Hale G, Gorus F, Goldman M, Walter M, Candon S, Schandene L, Crenier L, De Block C, Seigneurin JM, De Pauw P, Pierard D, Weets I, Rebello P, Bird P, Berrie E, Frewin M, Waldmann H, Bach JF, Pipeleers D, Chatenoud L. Insulin needs after CD3-antibody therapy in new-onset type 1 diabetes. N Engl J Med. 2005 Jun 23;352(25):2598-608. doi: 10.1056/NEJMoa043980. PMID 15972866
- [Background] You S, Candon S, Kuhn C, Bach JF, Chatenoud L. CD3 antibodies as unique tools to restore self-tolerance in established autoimmunity their mode of action and clinical application in type 1 diabetes. Adv Immunol. 2008;100:13-37. doi: 10.1016/S0065-2776(08)00802-X. No abstract available. PMID 19111162
- See also: Website containing information on DEFEND study — http://www.defendagainstdiabetes.com/
- Available data/document: Clinical Study Report: 115495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 85 centers in 9 countries namely Canada (4), Germany (3), Denmark (1), Spain (5), Finland (2), United Kingdom (4), Italy (8), Sweden (11) and United States of America (47) from 29 July 2008 to 31 January 2012. A total of 240 participants with new-onset Type 1 diabetes mellitus (NOT1DM) were planned to be enrolled.
Pre-assignment Details: Participants were screened for a period of 35 days and a total of 272 participants were randomized in the study.
Groups:
- Adolescent (Placebo): Eligible adolescent participants received matching placebo to Otelixizumab administered as intravenous (IV) infusions, with each infusion given over a 30-minute period. Participants received a series of 8 infusions, 1 infusion per Day over 8 consecutive days. Participants were followed-up for 24 months after the last dose.
- Adolescent (Otelixizumab): Eligible adolescent participants received Otelixizumab administered as IV infusions, with each infusion given over a 30-minute period. Participants received a series of 8 infusions as first dose (Day 1 of 0.1 milligram [mg], second dose (Day 2 of 0.2 mg), third dose (Day 3 of 0.3 mg), fourth, fifth, sixth, seventh and eight dose (on Days 4,5,6,7,8 of 0.5 mg per Day) 1 infusion per Day over 8 consecutive days . The total amount of Otelixizumab administered was 3.1 mg. Participants were followed-up for 24 months after the last dose.
- Adult (Placebo): Eligible adult participants received matching placebo to Otelixizumab administered as IV infusions, with each infusion given over a 30-minute period. Participants received a series of 8 infusions, 1 infusion per day over 8 consecutive Days. Participants were followed-up for 24 months after the last dose.
- Adult (Otelixizumab): Eligible adult participants received Otelixizumab administered as IV infusions, with each infusion given over a 30-minute period. Participants received a series of 8 infusions as first dose (Day 1 of 0.1 mg), second dose (Day 2 of 0.2 mg), third dose (Day 3 of 0.3 mg), fourth, fifth, sixth, seventh and eight dose (on Days 4,5,6,7,8 of 0.5 mg per Day) 1 infusion per Day over 8 consecutive days . The total amount of Otelixizumab administered was 3.1 mg. Participants were followed-up for 24 months after the last dose.
Period: Overall Study
Arm/Group | Adolescent (Placebo) | Adolescent (Otelixizumab) | Adult (Placebo) | Adult (Otelixizumab)
Started | 10 | 19 | 81 | 162
Completed | 10 | 19 | 72 | 153
Not Completed | 0 | 0 | 9 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 6
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants received matching placebo to Otelixizumab administered as IV infusions, with each infusion given over a 30-minute period. Participants received a series of 8 infusions, 1 infusion per Day over 8 consecutive days. Participants were followed-up for 24 months after the last dose.
- Otelixizumab: Eligible participants received Otelixizumab administered as IV infusions, with each infusion given over a 30-minute period. Participants received a series of 8 infusions as first dose (Day 1 of 0.1 mg, second dose (Day 2 of 0.2 mg), third dose (Day 3 of 0.3 mg), fourth, fifth, sixth, seventh and eight dose (on Days 4,5,6,7,8 of 0.5 mg per Day) 1 infusion per Day over 8 consecutive days . The total amount of Otelixizumab administered was 3.1 mg. Participants were followed-up for 24 months after the last dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Otelixizumab | Total
Number analyzed (Participants) | 91 | 181 | 272
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.2 (7.13) | 24.7 (6.54) | 24.9 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 64 | 95
  Male | 60 | 117 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 85 | 169 | 254
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 2-hour Mixed Meal Stimulated C-peptide Area Under Curve [AUC] (Normalized for 120-minute Time Interval) at Month 12
Description: Mixed meal-stimulated C-peptide AUC was the area under the C-peptide/time curve from Time 0 to 120 minutes, calculated using the trapezoidal rule. This reported AUC was normalized for time interval by dividing it by 120 minutes. This normalized AUC was calculated for each participant at Baseline, Week 12, and at Months 6, 12, 18, and 24. Data has been presented for meal stimulated C-peptide Area under assessment performed at Month 12. Baseline assessments were carried out on the morning of Day 1, before the start of the first infusion of study drug. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at Month 12.
Time Frame: Baseline (0-120 minutes on Day 1) and Month 12 (0-120 minutes)
Population: Intent-to-treat (ITT) population, comprised of all participants who were randomized and received any part of at least 1 infusion of study drug.
Measure: Least Squares Mean (Standard Error); unit: nanomoles per liter
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
nanomoles per liter | -0.21 (0.030) | -0.21 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Mixed meal-stimulated C-peptide AUC, Placebo Vs Otelixizumab at Month 12; Test type: Superiority or Other; p = 0.813, Mixed effects repeated measures model; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.06 to 0.08]

2. Secondary Outcome: Number of Participants Who Were Responders for (Glycosylated Hemoglobin) HbA1c/Insulin Use Response at Week 12 and Months 6 and 12
Description: A participant was considered a responder if, at the given time point, the participant had HbA1c<= 6.5%, and mean daily insulin use over 7 consecutive days < 0.5 international units per kilogram per day (IU/kg/day) during the 2 weeks preceding the visit. Data has been presented from number of participants with their percentages who were responders at Week 12 and Months 6 and 12.
Time Frame: Week 12 and Months 6 and 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Participants
  Responders at Week 12: number analyzed (Participants) | 78 | 161
  Responders at Week 12 | 45 | 85
  Responders at Month 6: number analyzed (Participants) | 76 | 158
  Responders at Month 6 | 42 | 74
  Responders at Month 12: number analyzed (Participants) | 80 | 160
  Responders at Month 12 | 34 | 56
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Percentage of responders, Placebo Vs Otelixizumab at Week 12; Test type: Superiority or Other; p = 0.737, Hochberg adjusted; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.47 to 1.70]
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Percentage of responders, Placebo Vs Otelixizumab at Month 6; Test type: Superiority or Other; p = 0.737, Hochberg adjusted; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.42 to 1.39]
Statistical Analysis 3: Comparison: Placebo vs Otelixizumab; Percentage of responders, Placebo Vs Otelixizumab at Month 12; Test type: Superiority or Other; p = 0.481, Hochberg adjusted; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.45 to 1.46]

3. Secondary Outcome: Mean Daily Insulin Use at Week 12 and Months 6 and 12.
Description: Participants recorded their daily insulin use in their electronic diaries. In particular, insulin was recorded thoroughly and accurately for at least 7 consecutive days during the 2 weeks before the visits at Baseline, Week 12, and Months 6 and 12. During each of these visits, the investigator/designee accessed the invivodata DiaryPRO web site to review insulin-use data for the previous 2-week period to ensure completeness. If errors/gaps were identified (e.g., if the participant did not take insulin and not entered 0 units), the investigator/designee recorded the missing data from participant recall using a data clarification form (DCF). Paper diary to collect insulin use, were reviewed for completeness. Any missing data that could be recalled by the participant was entered. If the participant did not record any insulin use during the 2-week period before the visit, the site obtained an insulin use history for the previous 7 days and calculated the average daily insulin dose.
Time Frame: Week 12 and Months 6 and 12.
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: IU/kg
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
IU/kg
  Mean daily insulin use at Week 12 | 0.34 (0.017) | 0.31 (0.013)
  Mean daily insulin use at Month 6 | 0.36 (0.022) | 0.36 (0.016)
  Mean daily insulin use at Month 12 | 0.42 (0.023) | 0.39 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Mean insulin use, Placebo Vs Otelixizumab at Week 12; Test type: Superiority or Other; p = 0.281, Mixed effects repeated measures model; Mixed effects repeated measures models was adjusted for age, continent, and baseline parameter value; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.07 to 0.01]
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Mean insulin use, Placebo Vs Otelixizumab at Month 6; Test type: Superiority; p = 0.969, Mixed effects repeated measures model; Mixed effects repeated measures models was adjusted for age, continent, and baseline parameter value; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.05 to 0.05]
Statistical Analysis 3: Comparison: Placebo vs Otelixizumab; Mean insulin use, Placebo Vs Otelixizumab at Month 12; Test type: Superiority or Other; p = 0.272, Mixed effects repeated measures model; Mixed effects repeated measures models was adjusted for age, continent, and baseline parameter value; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.08 to 0.02]

4. Secondary Outcome: HbA1c Level at Week 12 and Months 6 and 12
Description: HbA1c levels were recorded at Screening, Baseline (Day 1), Day 28, Week 8, Week 12, Months 4 to 12 and Month 24. Data has been presented for HbA1c levels at Week 12 and Months 6 and 12.
Time Frame: Week 12 and Months 6 and 12
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Percentage
  HbA1c levels at Month 12 | 6.83 (0.146) | 7.02 (0.108)
  HbA1c levels at Month 6 | 6.60 (0.138) | 6.77 (0.100)
  HbA1c levels at Week 12 | 6.45 (0.124) | 6.54 (0.094)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; HbA1c levels, Placebo Vs Otelixizumab at Month 12; Test type: Superiority or Other; p = 0.289, Mixed effects repeated measures model; Mixed effects repeated measures models was adjusted for age, continent, and baseline parameter value; Median Difference (Final Values) = 0.18, 95% CI 2-sided [-0.16 to 0.52]
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; HbA1c levels, Placebo Vs Otelixizumab at Month 6; Test type: Superiority or Other; p = 0.538, Mixed effects repeated measures model; Mixed effects repeated measures models was adjusted for age, continent, and baseline parameter value; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.15 to 0.49]
Statistical Analysis 3: Comparison: Placebo vs Otelixizumab; HbA1c levels, Placebo Vs Otelixizumab at Week 12; Test type: Superiority or Other; p = 0.538, Mixed effects repeated measures model; Mixed effects repeated measures models was adjusted for age, continent, and baseline parameter value; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.19 to 0.36]

5. Secondary Outcome: Number of Hypoglycemic Events Defined by Hypoglycemic Event Categories From Baseline Upto Month 12
Description: Hypoglycemic events reported by participants were classified as defined by the American Diabetes Association (ADA) Workgroup on Hypoglycemia as follows: Severe hypoglycemia: an event requiring assistance of another person to actively administer carbohydrate, glucagon/other resuscitative actions, documented symptomatic hypoglycemia: an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration(PGC)<=70 mg/dL, asymptomatic hypoglycemia: an event not accompanied by typical symptoms of hypoglycemia but with a measured PGC<=70 mg/dL,probable symptomatic hypoglycemia: an event during which symptoms of hypoglycemia are not accompanied by a plasma glucose determination, but were presumably caused by a PGC<=70 mg/dL and relative hypoglycemia: an event during which the person with diabetes reports any of the typical symptoms of hypoglycemia, and interprets the symptoms as indicative of hypoglycemia, but with a measured PGC>70 mg/dL.
Time Frame: Upto Month 12
Population: ITT population.
Measure: Number; unit: Hypoglycemic events
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Hypoglycemic events
  Severe hypoglycemia upto Month 12 | 2 | 5
  Documented symptomatic hypoglycemia upto Month 12 | 3092 | 6322
  Asymptomatic hypoglycemia upto Month 12 | 4718 | 9962
  Probable symptomatic hypoglycemia upto Month 12 | 84 | 93
  Relative hypoglycemia upto Month 12 | 85 | 211

6. Secondary Outcome: Number of Participants With Hypoglycemic Events Defined by Hypoglycemic Event Categories From Baseline Upto Month 12
Description: Hypoglycemic events reported by participants were classified as defined by the ADA Workgroup on Hypoglycemia as Severe hypoglycemia: an event requiring assistance of another person to actively administer carbohydrate, glucagon/other resuscitative actions, documented symptomatic hypoglycemia: an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration (PGC)<=70 mg/dL, asymptomatic hypoglycemia: an event not accompanied by typical symptoms of hypoglycemia but with a measured PGC<=70 mg/dL,probable symptomatic hypoglycemia: an event during which symptoms of hypoglycemia are not accompanied by a plasma glucose determination, but were presumably caused by a PGC<=70 mg/dL and relative hypoglycemia: an event during which the person with diabetes reports any of the typical symptoms of hypoglycemia, and interprets the symptoms as indicative of hypoglycemia, but with a measured PGC>70 mg/dL. Only categories with values are presented.
Time Frame: Upto Month 12
Population: ITT population. Data has been presented for number of participants with their percentages with hypoglycemic events defined by hypoglycemic event categories from Baseline upto month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Participants
  Severe hypoglycemia upto Month 12 | 2 | 4
  Documented symptomatic hypoglycemia upto Month 12 | 78 | 163
  Asymptomatic hypoglycemia upto Month 12 | 10 | 13

7. Secondary Outcome: Number of Hypoglycemic Excursions (<=70 mg/dL) With Most Complete Glucose at Week 12 and Months 6 and 12.
Description: The event frequency of glucose measurements that were hypoglycemic excursions were calculated per participant basis, using the number of occurrences where blood glucose was less than or equal to 70 mg/dL. Most complete glucose interval was the 7 day period with the maximum number of days with at least 4 recordings per day. If these results were in more than one 7 day period, then the 7 day period with the largest average number of daily recordings (out of those with the maximum number of days with at least 4 recordings per day) was selected. If there were 2 or more 7 day periods that have the same number of days with at least 4 recordings and the same maximum average number of glucose recordings, the period that ended closest to the day of the study was selected.
Time Frame: Week 12 and Months 6 and 12.
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Hypoglycemic excursions
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Hypoglycemic excursions
  Number of hypoglycemic excursions at Week 12: number analyzed (Participants) | 90 | 177
  Number of hypoglycemic excursions at Week 12 | 2.3 (0.28) | 2.8 (0.27)
  Number of hypoglycemic excursions at Month 6: number analyzed (Participants) | 80 | 166
  Number of hypoglycemic excursions at Month 6 | 3.0 (0.36) | 2.9 (0.27)
  Number of hypoglycemic excursions at Month 12: number analyzed (Participants) | 78 | 161
  Number of hypoglycemic excursions at Month 12 | 2.9 (0.41) | 3.2 (0.32)

8. Secondary Outcome: Magnitude of Greatest Hypoglycemic Excursions With Most Complete Glucose at Week 12 and Months 6 and 12.
Description: The greatest hypoglycemic excursions during an interval was calculated as 70 mg/dL minus the lowest recorded glucose level in the interval. If a participant had data recorded during the interval but did not have a value below 70 mg/dL, the participants greatest hypoglycemic excursion for that interval was 0 mg/dL.
  Most complete glucose interval was the 7 day period with the maximum number of days with at least 4 recordings per day. If these results were in more than one 7 day period, then the 7 day period with the largest average number of daily recordings (out of those with the maximum number of days with at least 4 recordings per day) was selected. If there were 2 or more 7 day periods that have the same number of days with at least 4 recordings and the same maximum average number of glucose recordings, the period that ended closest to the day of the study was selected.
Time Frame: Week 12 and Months 6 and 12.
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: milligrams per deciliter
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
milligrams per deciliter
  Magnitude of excursion, Week 12: number analyzed (Participants) | 90 | 177
  Magnitude of excursion, Week 12 | 9.4 (0.92) | 10.8 (0.90)
  Magnitude of excursion, Month 6: number analyzed (Participants) | 80 | 166
  Magnitude of excursion, Month 6 | 11.9 (1.24) | 10.6 (0.77)
  Magnitude of excursion, Month 12: number analyzed (Participants) | 78 | 161
  Magnitude of excursion, Month 12 | 11.2 (1.20) | 11.0 (0.92)

9. Secondary Outcome: Number of Participants With Hypoglycemic Excursions With Most Complete Glucose at Week 12 and Months 6 and 12
Description: Percentage of hypoglycemic excursions was calculated as the total number of observations that exceed the hypoglycemic excursion boundary (i.e.<= 70 mg/dL) divided by the total number of glucose measurements recorded in a time interval for the intervals: Baseline to Week 12, post-Week 12 to Month 6, post-Month 6 to Month 12. Most complete glucose interval was the 7 day period with the maximum number of days with at least 4 recordings per day. If these results were in more than one 7 day period, then the 7 day period with the largest average number of daily recordings (out of those with the maximum number of days with at least 4 recordings per day) was selected. If there were 2 or more 7 day periods that have the same number of days with at least 4 recordings and the same maximum average number of glucose recordings, the period that ended closest to the day of the study was selected. Data has been presented for number of participants with their percentages having hypoglycemic excursion.
Time Frame: Week 12 and Months 6 and 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Participants
  Percentage of participants with excursion,Week 12: number analyzed (Participants) | 90 | 177
  Percentage of participants with excursion,Week 12 | 72 | 127
  Percentage of participants with excursion,Month 6: number analyzed (Participants) | 80 | 166
  Percentage of participants with excursion,Month 6 | 57 | 121
  Percentage of participants with excursion,Month 12: number analyzed (Participants) | 78 | 161
  Percentage of participants with excursion,Month 12 | 56 | 111

10. Secondary Outcome: Number of Hyperglycemic Excursions With Most Complete Glucose at Week 12 and Months 6 and 12.
Description: The event frequency of glucose measurements that were hyperglycemic excursions were calculated on a per participant basis using the number of occurrences where blood glucose was greater than the hyperglycemic tolerance limit. There were 3 hyperglycemic tolerance limits considered: 200 mg/dL, 130 mg/dL and 100 mg/dL. Most complete glucose interval was the 7 day period with the maximum number of days with at least 4 recordings per day. If these results were in more than one 7 day period, then the 7 day period with the largest average number of daily recordings (out of those with the maximum number of days with at least 4 recordings per day) was selected. If there were 2 or more 7 day periods that have the same number of days with at least 4 recordings and the same maximum average number of glucose recordings, the period that ended closest to the day of the study was selected.
Time Frame: Week 12 and Months 6 and 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Hyperglycemic excursions
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Hyperglycemic excursions
  Threshold > 100 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold > 100 mg/dL at Week 12 | 34.0 (1.78) | 32.9 (1.15)
  Threshold > 130 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold > 130 mg/dL at Week 12 | 20.5 (1.72) | 19.9 (1.01)
  Threshold > 200 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold > 200 mg/dL at Week 12 | 5.7 (0.85) | 5.6 (0.59)
  Threshold > 100 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold > 100 mg/dL at Month 6 | 33.5 (1.77) | 35.1 (1.41)
  Threshold > 130 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold > 130 mg/dL at Month 6 | 20.8 (1.68) | 22.7 (1.25)
  Threshold > 200 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold > 200 mg/dL at Month 6 | 6.5 (1.07) | 7.9 (0.85)
  Threshold > 100 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold > 100 mg/dL at Month 12 | 35.6 (1.97) | 33.4 (1.27)
  Threshold > 130 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold > 130 mg/dL at Month 12 | 24.0 (1.92) | 22.2 (1.05)
  Threshold > 200 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold > 200 mg/dL at Month 12 | 8.6 (1.42) | 6.9 (0.59)

11. Secondary Outcome: Magnitude of Greatest Hyperglycemic Excursions With Most Complete Glucose at Week 12 and Months 6 and 12.
Description: The greatest hyperglycemic excursions during an interval was calculated as the largest recorded glucose level in the interval minus the hyperglycemic tolerance limit value (HGTLV). If a participant had data recorded during the interval but did not have a value above the HGTLV, the participants greatest hyperglycemic excursion for that interval was 0 mg/dL. Most complete glucose interval was the 7 day period with the maximum number of days with at least 4 recordings per day. If these results were in more than one 7 day period, then the 7 day period with the largest average number of daily recordings (out of those with the maximum number of days with at least 4 recordings per day) was selected. If there were 2 or more 7 day periods that have the same number of days with at least 4 recordings and the same maximum average number of glucose recordings, the period that ended closest to the day of the study was selected.
Time Frame: Week 12 and Months 6 and 12.
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: milligrams per deciliter
Groups:
- Placebo: Eligible participants received matching placebo to Otelixizumab administered as IV infusions, with each infusion given over a 30-minute period. Participants received a series of 8 infusions, 1 infusion per day over 8 consecutive days.
- Otelixizumab: Eligible participants received Otelixizumab administered as IV infusions, with each infusion given over a 30-minute period. Participants received a series of 8 infusions (as first dose-day 1 of 0.1 mg, second dose-day 2 of 0.2 mg, third dose-day 3 of 0.3 mg, fourth, fifth, sixth, seventh and eight dose on days 4,5,6,7,8 of 0.5 mg per day) 1 infusion per day over 8 consecutive days . The total amount of Otelixizumab administered was 3.1 mg.
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
milligrams per deciliter
  Threshold> 100 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold> 100 mg/dL at Week 12 | 158.3 (9.26) | 158.4 (6.65)
  Threshold> 130 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold> 130 mg/dL at Week 12 | 128.3 (9.26) | 128.4 (6.65)
  Threshold> 200 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold> 200 mg/dL at Week 12 | 65.7 (8.51) | 65.7 (6.12)
  Threshold> 100 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold> 100 mg/dL at Month 6 | 154.6 (9.34) | 175.7 (8.09)
  Threshold> 130 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold> 130 mg/dL at Month 6 | 124.8 (9.31) | 145.7 (8.09)
  Threshold> 200 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold> 200 mg/dL at Month 6 | 63.3 (8.32) | 80.1 (7.75)
  Threshold> 100 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold> 100 mg/dL at Month 12 | 176.7 (10.02) | 177.5 (7.08)
  Threshold> 130 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold> 130 mg/dL at Month 12 | 146.8 (10.00) | 147.5 (7.07)
  Threshold> 200 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold> 200 mg/dL at Month 12 | 81.8 (9.33) | 82.6 (6.61)

12. Secondary Outcome: Number of Participants With Hyperglycemic Excursions With Most Complete Glucose at Week 12 and Months 6 and 12
Description: Percentage of hyperglycemic excursions was calculated as the total number of observations that exceed the hyperglycemic excursion boundary (i.e. > HGTLV) divided by the total number of glucose measurements recorded in a time interval for the intervals: Baseline to Week 12, post-Week 12 to Month 6, post-Month 6 to Month 12. Most complete glucose interval was the 7 day period with the maximum number of days with at least 4 recordings per day. If these results were in more than one 7 day period, then the 7 day period with the largest average number of daily recordings (out of those with the maximum number of days with at least 4 recordings per day) was selected. If there were 2 or more 7 day periods that have the same number of days with at least 4 recordings and the same maximum average number of glucose recordings, the period that ended closest to the day of the study was selected. Data for number of participants with their percentages are presented.
Time Frame: Week 12 and Months 6 and 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Participants
  Threshold> 100 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold> 100 mg/dL at Week 12 | 90 | 177
  Threshold> 130 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold> 130 mg/dL at Week 12 | 90 | 177
  Threshold> 200 mg/dL at Week 12: number analyzed (Participants) | 90 | 177
  Threshold> 200 mg/dL at Week 12 | 65 | 130
  Threshold> 100 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold> 100 mg/dL at Month 6 | 80 | 166
  Threshold> 130 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold> 130 mg/dL at Month 6 | 79 | 166
  Threshold> 200 mg/dL at Month 6: number analyzed (Participants) | 80 | 166
  Threshold> 200 mg/dL at Month 6 | 57 | 139
  Threshold> 100 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold> 100 mg/dL at Month 12 | 78 | 161
  Threshold> 130 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold> 130 mg/dL at Month 12 | 77 | 160
  Threshold> 200 mg/dL at Month 12: number analyzed (Participants) | 78 | 161
  Threshold> 200 mg/dL at Month 12 | 60 | 131

13. Secondary Outcome: Change From Baseline in Average Daily Risk Range (ADRR) at Week 12 and Months 6 and 12.
Description: Average daily risk range is a measure for evaluation of blood glucose variability that was designed to be equally sensitive to hypoglycemia and hyperglycemia. The ADRR was assessed over 30-day periods prior to Baseline and at key visits Week 12 and Months 6 and 12. Baseline assessments were carried out on the morning of Day 1, before the start of the first infusion of study drug. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at Week 12 and Months 6 and 12.
Time Frame: Baseline (Day 1) and Week 12, Months 6 and 12.
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Ratio
  ADRR at Week 12 | -0.41 (0.826) | 0.71 (0.599)
  ADRR at Month 6 | 2.03 (1.133) | 2.86 (0.801)
  ADRR at Month 12 | 3.29 (1.038) | 4.22 (0.732)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; ADRR, Placebo Vs Otelixizumab at Week 12; Test type: Superiority or Other; p = 0.540, Mixed effects repeated measures model; Median Difference (Net) = 1.12, 95% CI 2-sided [-0.88 to 3.11]
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; ADRR, Placebo Vs Otelixizumab at Month 6; Test type: Superiority or Other; p = 0.546, Mixed effects repeated measures model; Mean Difference (Net) = 0.83, 95% CI 2-sided [-1.89 to 3.56]
Statistical Analysis 3: Comparison: Placebo vs Otelixizumab; ADRR, Placebo Vs Otelixizumab at Month 12; Test type: Superiority or Other; p = 0.462, Mixed effects repeated measures model; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-1.56 to 3.42]

14. Secondary Outcome: Composite Rank Summary for HbA1c and Exogenous Insulin Use at Month 6 and Month 12
Description: O'Brien mean rank analyses was performed on a two-part composite of the baseline-adjusted HbA1c level and the baseline-adjusted mean total daily insulin use per kg body weight in the otelixizumab group compared with the placebo group at Months 6, 12. For the O'Brien mean rank analysis at a particular time point, adjusted HbA1c values (for both treatment groups together) was ranked from smallest to largest, and adjusted mean daily insulin use values were ranked from smallest to largest. For each participant, the HbA1c and insulin use ranks were added together, producing a composite rank. A treatment comparison test was then performed on the composite ranks.
Time Frame: Month 6 and 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Composite rank score
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Composite rank score
  Composite rank summary, Month 6: number analyzed (Participants) | 73 | 156
  Composite rank summary, Month 6 | 238 (123.3) | 247 (113.7)
  Composite rank summary, Month 12: number analyzed (Participants) | 76 | 158
  Composite rank summary, Month 12 | 245 (120.0) | 244 (115.2)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Composite Rank Summary for HbA1c and Exogenous Insulin Use, Placebo Vs Otelixizumab at Month 6; Test type: Superiority or Other; p = 0.957, Hochberg-adjusted
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Composite Rank Summary for HbA1c and Exogenous Insulin Use, Placebo Vs Otelixizumab at Month 12; Test type: Superiority or Other; p = 0.957, Hochberg-adjusted

15. Secondary Outcome: Composite Rank Summary for C-Peptide AUC, HbA1c and Exogenous Insulin Use at Month 6 and Month 12
Description: O'Brien analyses will be performed on a three-part composite of HbA1c level, C-peptide AUC, and mean daily Insulin use in the otelixizumab group compared with the placebo group at Months 6 and12. For the O'Brien mean rank analysis at a particular time point, HbA1c and insulin use will be ranked from smallest to largest, and C-peptide AUC will be ranked from largest to smallest. For each participant, the C-Peptide AUC, ranks for HbA1c and insulin use were added together, producing a composite rank. A treatment comparison test was then performed on the composite ranks.
Time Frame: Month 6 and 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Composite rank score
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Composite rank score
  Month 6: number analyzed (Participants) | 72 | 151
  Month 6 | 365 (83.8) | 373 (105.6)
  Month 12: number analyzed (Participants) | 74 | 151
  Month 12 | 360 (85.1) | 366 (95.4)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Composite Rank Summary for C-Peptide AUC, HbA1c and Exogenous Insulin Use, Placebo Vs Otelixizumab at Month 6; Test type: Superiority or Other; p = 0.653, Hochberg-adjusted
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Composite Rank Summary for C-Peptide AUC, HbA1c and Exogenous Insulin Use, Placebo Vs Otelixizumab at Month 12; Test type: Superiority or Other; p = 0.653, Hochberg-adjusted

16. Secondary Outcome: Change From Baseline in Level of Cytokines Interleukin (IL-6), IL-10 and Tumor Necrosis Factor-alpha (TNF-a) at Day 1, Day 4, Day 8
Description: Levels of cytokine (TNFα, IL-6, IL-10) were measured at Baseline and at 2 hours after end of infusion (EOI) on Day 1, Day 4, Day 8 . Baseline assessments were carried out on the morning of Day 1, before the start of the first infusion of study drug. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at Day 1, Day 4 and Day 8.
Time Frame: Day 1, Day 4, Day 8
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: picograms per milliliter
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
picograms per milliliter
  IL-6 levels, Day 1, 2 hours after EOI: number analyzed (Participants) | 24 | 50
  IL-6 levels, Day 1, 2 hours after EOI | 0.76 (0.680) | 2.78 (0.544)
  IL-6 levels, Day 4, 2 hours after EOI: number analyzed (Participants) | 24 | 44
  IL-6 levels, Day 4, 2 hours after EOI | -0.13 (0.251) | 3.01 (1.107)
  IL-6 levels, Day 8, 2 hours after EOI: number analyzed (Participants) | 23 | 50
  IL-6 levels, Day 8, 2 hours after EOI | 0.45 (0.448) | 14.59 (5.266)
  IL-10 levels, Day 1, 2 hours after EOI: number analyzed (Participants) | 23 | 50
  IL-10 levels, Day 1, 2 hours after EOI | 0.15 (0.342) | 4.61 (1.770)
  IL-10 levels, Day 4, 2 hours after EOI: number analyzed (Participants) | 23 | 44
  IL-10 levels, Day 4, 2 hours after EOI | 0.55 (0.629) | 1.35 (0.575)
  IL-10 levels, Day 8, 2 hours after EOI: number analyzed (Participants) | 22 | 49
  IL-10 levels, Day 8, 2 hours after EOI | 1.84 (1.019) | 25.57 (7.196)
  TNF-a levels, Day 1, 2 hours after EOI: number analyzed (Participants) | 24 | 50
  TNF-a levels, Day 1, 2 hours after EOI | -0.126 (0.0719) | 2.320 (0.3996)
  TNF-a levels, Day 4, 2 hours after EOI: number analyzed (Participants) | 24 | 44
  TNF-a levels, Day 4, 2 hours after EOI | 0.111 (0.2381) | 1.509 (0.5740)
  TNF-a levels, Day 8, 2 hours after EOI: number analyzed (Participants) | 23 | 50
  TNF-a levels, Day 8, 2 hours after EOI | 0.135 (0.2649) | 3.614 (0.8920)

17. Secondary Outcome: Percent Change From Baseline in Circulating Peripheral Lymphocytes CD4+CD25+FoxP3+ T Cells and CD4+CD25hiFoxP3+ T Cells in Type 1 Diabetes Mellitus (TIDM) up to Month 12
Description: Blood samples were drawn for lymphocyte subset evaluations at Baseline and at 2hours after EOI on Day 4, pre-dose and after E0I on Day 8, Day 14, Day 21, Day 28, Week 6, Week 8, Week 10, Week 12, Month 6 and Month 12. Percentages of relevant lymphocyte subsets were determined by flow cytometry. The lymphocyte subsets assessed included CD8+CD25+ T lymphocytes, as well as the subsets of lymphocytes of these type that were positive for FoxP3, a protein that was expressed at high levels in the cytoplasm of regulatory T cells. CD4+CD25hiFoxP3+ T lymphocytes, a cell type was of interest because it played a regulatory role in T1DM. Baseline assessments were carried out on the morning of Day 1, before the start of the first infusion of study drug. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (pre-dose on Day 1) and up to 12 Months
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Percent change
  CD4+CD25+FoxP3+ T, Day 4, 2 hours after EOI: number analyzed (Participants) | 28 | 56
  CD4+CD25+FoxP3+ T, Day 4, 2 hours after EOI | 118.8 [32.1 to 366.9] | 53.4 [3.4 to 235.9]
  CD4+CD25+FoxP3+ T, Day 8 pre-dose: number analyzed (Participants) | 27 | 57
  CD4+CD25+FoxP3+ T, Day 8 pre-dose | 94.4 [25.9 to 199.9] | 49.7 [9.4 to 148.5]
  CD4+CD25+FoxP3+ T, Day 8, 2 hours after EOI: number analyzed (Participants) | 70 | 146
  CD4+CD25+FoxP3+ T, Day 8, 2 hours after EOI | 113.2 [28.8 to 2127.6] | 40.1 [2.1 to 3737.0]
  CD4+CD25+FoxP3+ T, Day 14: number analyzed (Participants) | 72 | 153
  CD4+CD25+FoxP3+ T, Day 14 | 114.5 [26.5 to 2384.4] | 101.3 [15.5 to 10906.4]
  CD4+CD25+FoxP3+ T, Day 21: number analyzed (Participants) | 74 | 147
  CD4+CD25+FoxP3+ T, Day 21 | 114.6 [34.8 to 489.8] | 101.9 [0.0 to 44228.1]
  CD4+CD25+FoxP3+ T, Day 28: number analyzed (Participants) | 75 | 151
  CD4+CD25+FoxP3+ T, Day 28 | 95.1 [7.0 to 1612.7] | 101.7 [2.1 to 6363.7]
  CD4+CD25+FoxP3+ T, Week 6: number analyzed (Participants) | 72 | 148
  CD4+CD25+FoxP3+ T, Week 6 | 104.1 [0.0 to 514.2] | 106.6 [0.0 to 7010.9]
  CD4+CD25+FoxP3+ T, Week 8: number analyzed (Participants) | 75 | 156
  CD4+CD25+FoxP3+ T, Week 8 | 110.1 [29.1 to 1602.3] | 107.1 [4.7 to 15806.4]
  CD4+CD25+FoxP3+ T, Week 10: number analyzed (Participants) | 75 | 145
  CD4+CD25+FoxP3+ T, Week 10 | 109.9 [8.6 to 1820.9] | 102.7 [7.4 to 9943.6]
  CD4+CD25+FoxP3+ T, Week 12: number analyzed (Participants) | 75 | 150
  CD4+CD25+FoxP3+ T, Week 12 | 102.5 [9.8 to 1018.7] | 85.5 [2.9 to 9911.7]
  CD4+CD25+FoxP3+ T, Month 6: number analyzed (Participants) | 72 | 146
  CD4+CD25+FoxP3+ T, Month 6 | 137.9 [19.5 to 1409.6] | 133.3 [19.8 to 10357.4]
  CD4+CD25+FoxP3+ T, Month 12: number analyzed (Participants) | 70 | 149
  CD4+CD25+FoxP3+ T, Month 12 | 122.0 [9.5 to 628.7] | 106.9 [0.4 to 31690.3]
  CD4+CD25hiFoxP3+ T Cells, Day 4, 2 hours after EOI: number analyzed (Participants) | 28 | 56
  CD4+CD25hiFoxP3+ T Cells, Day 4, 2 hours after EOI | 151.9 [12.6 to 400.8] | 60.8 [1.5 to 364.5]
  CD4+CD25hiFoxP3+ T Cells, Day 8 pre-dose: number analyzed (Participants) | 27 | 57
  CD4+CD25hiFoxP3+ T Cells, Day 8 pre-dose | 93.8 [13.6 to 521.7] | 43.5 [3.6 to 675.0]
  CD4+CD25hiFoxP3+ T Cells, Day 8, 2 hours after EOI: number analyzed (Participants) | 69 | 146
  CD4+CD25hiFoxP3+ T Cells, Day 8, 2 hours after EOI | 110.7 [18.6 to 3577.8] | 35.9 [0.0 to 321279]
  CD4+CD25hiFoxP3+ T Cells, Day 14: number analyzed (Participants) | 71 | 153
  CD4+CD25hiFoxP3+ T Cells, Day 14 | 118.4 [8.8 to 1502.5] | 109.7 [5.8 to 1364664]
  CD4+CD25hiFoxP3+ T Cells, Day 21: number analyzed (Participants) | 74 | 147
  CD4+CD25hiFoxP3+ T Cells, Day 21 | 110.0 [9.7 to 1720.2] | 98.8 [0.0 to 1479653]
  CD4+CD25hiFoxP3+ T Cells, Day 28: number analyzed (Participants) | 74 | 151
  CD4+CD25hiFoxP3+ T Cells, Day 28 | 101.1 [2.1 to 949.9] | 108.7 [0.0 to 62190.9]
  CD4+CD25hiFoxP3+ T Cells, Week 6: number analyzed (Participants) | 72 | 148
  CD4+CD25hiFoxP3+ T Cells, Week 6 | 106.9 [0.0 to 2508.7] | 110.7 [0.0 to 9573.5]
  CD4+CD25hiFoxP3+ T Cells, Week 8: number analyzed (Participants) | 74 | 156
  CD4+CD25hiFoxP3+ T Cells, Week 8 | 131.7 [14.1 to 843.2] | 120.3 [0.5 to 175040]
  CD4+CD25hiFoxP3+ T Cells, Week 10: number analyzed (Participants) | 74 | 145
  CD4+CD25hiFoxP3+ T Cells, Week 10 | 97.7 [1.5 to 2356.8] | 107.0 [0.0 to 128591]
  CD4+CD25hiFoxP3+ T Cells, Week 12: number analyzed (Participants) | 74 | 150
  CD4+CD25hiFoxP3+ T Cells, Week 12 | 113.6 [1.9 to 1310.2] | 90.9 [0.1 to 1045228]
  CD4+CD25hiFoxP3+ T Cells, Month 6: number analyzed (Participants) | 71 | 146
  CD4+CD25hiFoxP3+ T Cells, Month 6 | 150.9 [6.1 to 25639.5] | 153.2 [5.5 to 1544544]
  CD4+CD25hiFoxP3+ T Cells, Month 12: number analyzed (Participants) | 69 | 149
  CD4+CD25hiFoxP3+ T Cells, Month 12 | 166.4 [5.1 to 1748.9] | 160.6 [0.0 to 78843.4]

18. Secondary Outcome: Percent Change From Baseline in Cell-bound Otelixizumab on CD4+ T Cells at Day 1, Day 4, Day 8
Description: The amount of cell-bound otelixizumab was determined by flow cytometry. The extent of T cell receptor alpha beta (TCRαβ) expression was determined using an antibody that bound to TCRαβ but did not compete with otelixizumab for binding sites at the expected range of concentrations. The MESF of the anti-TCRαβ antibody was used to quantify the number of CD3/TCR complexes present on T cells. Free otelixizumab binding sites (sites not occupied by otelixizumab) were detected by staining with biotinylated otelixizumab. The MESF of bound biotinylated otelixizumab was directly proportional to the availability of free otelixizumab binding sites. MESF of bound antibody on CD4+ T cells was a direct measurement of cell-bound otelixizumab on CD4+ T cells. Baseline assessments were carried out on the morning of Day 1, before the start of the first infusion of study drug. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at Day 1, Day 4 and Day 8.
Time Frame: Baseline (pre-dose on Day 1), Day 4 and Day 8
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Percent change
  CD4+ T cells, Day 1, 2 hours after EOI: number analyzed (Participants) | 20 | 57
  CD4+ T cells, Day 1, 2 hours after EOI | 125.1 (18.00) | 914.8 (269.18)
  CD4+ T cells, Day 4, 2 hours after EOI: number analyzed (Participants) | 23 | 54
  CD4+ T cells, Day 4, 2 hours after EOI | 174.3 (41.95) | 2719.8 (369.41)
  CD4+ T cells, Day 8, pre-dose: number analyzed (Participants) | 26 | 54
  CD4+ T cells, Day 8, pre-dose | 151.5 (39.49) | 471.5 (98.53)
  CD4+ T cells, Day 8, 2 hours after EOI: number analyzed (Participants) | 26 | 57
  CD4+ T cells, Day 8, 2 hours after EOI | 167.9 (47.67) | 1387.5 (274.21)

19. Secondary Outcome: Percent Change From Baseline in CD3/TCR Saturation on CD4+ T Cells and CD8+ T Cells at Day 1, Day 4, Day 8
Description: The extent of saturation of CD3/TCR receptors on CD4+ and CD8+ lymphocytes was determined by flow cytometry. The extent of TCRαβ expression was determined using an antibody that bound to TCRαβ but did not compete with otelixizumab for binding sites at the expected range of concentrations. The MESF of the anti-TCRαβ antibody was used to quantify the number of CD3/TCR complexes present on T cells. The MESF of bound biotinylated otelixizumab was directly proportional to the availability of free otelixizumab binding sites. MESF of free CD3 sites on CD4+ T cells and CD8+ T cells was direct measurement of saturation of the CD3/TCR complex on CD4+ T cells and CD8+ T cells. Baseline assessments were carried out on the morning of Day 1, before the start of the first infusion of study drug. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at Day 1, Day 4 and Day 8.
Time Frame: Baseline (Pre-dose Day 1), Day 4, Day 8
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Percent change
  CD4+ T cells, Day 1, 2 hours after EOI: number analyzed (Participants) | 20 | 57
  CD4+ T cells, Day 1, 2 hours after EOI | 93.4 (2.40) | 90.9 (3.82)
  CD4+ T cells, Day 4, 2 hours after EOI: number analyzed (Participants) | 23 | 54
  CD4+ T cells, Day 4, 2 hours after EOI | 109.7 (11.91) | 50.2 (4.90)
  CD4+ T cells, Day 8, pre-dose: number analyzed (Participants) | 26 | 54
  CD4+ T cells, Day 8, pre-dose | 97.7 (10.66) | 59.0 (5.31)
  CD4+ T cells, Day 8, 2 hours after EOI: number analyzed (Participants) | 26 | 56
  CD4+ T cells, Day 8, 2 hours after EOI | 98.0 (13.03) | 21.7 (3.33)
  CD8+ T cells, Day 1, 2 hours after EOI: number analyzed (Participants) | 20 | 57
  CD8+ T cells, Day 1, 2 hours after EOI | 92.4 (2.38) | 91.4 (3.82)
  CD8+ T cells, Day 4, 2 hours after EOI: number analyzed (Participants) | 23 | 54
  CD8+ T cells, Day 4, 2 hours after EOI | 116.7 (14.53) | 51.6 (5.23)
  CD8+ T cells, Day 8, pre-dose: number analyzed (Participants) | 26 | 54
  CD8+ T cells, Day 8, pre-dose | 97.4 (11.84) | 60.8 (6.11)
  CD8+ T cells, Day 8, 2 hours after EOI: number analyzed (Participants) | 26 | 56
  CD8+ T cells, Day 8, 2 hours after EOI | 98.2 (14.63) | 23.0 (3.72)

20. Secondary Outcome: Percent Change From Baseline in CD3/TCR Modulation on CD4+ T Cells and CD8+ T Cells at Day 1, Day 4, Day 8
Description: The extent of modulation of CD3/TCR receptors on CD4+ and CD8+ lymphocytes was determined by flow cytometry. The extent of TCRαβ expression was determined using an antibody that bound to TCRαβ but did not compete with otelixizumab for binding sites at the expected range of concentrations. The MESF of the anti-TCRαβ antibody was used to quantify the number of CD3/TCR complexes present on T cells. The MESF of bound biotinylated otelixizumab was directly proportional to the availability of free otelixizumab binding sites.CD3/TCR complexes on CD4+ and CD8+ T cells were detected with a non-competing antibody. Changes in the MESF of TCR expression was a direct measurement of TCR modulation. Baseline assessments were carried out on the morning of Day 1, before the start of the first infusion of study drug. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at Day 1, Day 4 and Day 8.
Time Frame: Baseline (Pre-dose Day 1), Day 4, Day 8
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 91 | 181
Percent change
  CD4+ T cells, Day 1, 2 hours after EOI: number analyzed (Participants) | 20 | 57
  CD4+ T cells, Day 1, 2 hours after EOI | 94.2 (2.95) | 91.1 (2.90)
  CD4+ T cells, Day 4, 2 hours after EOI: number analyzed (Participants) | 23 | 54
  CD4+ T cells, Day 4, 2 hours after EOI | 103.8 (8.93) | 70.8 (3.89)
  CD4+ T cells, Day 8, pre-dose: number analyzed (Participants) | 26 | 54
  CD4+ T cells, Day 8, pre-dose | 101.4 (6.09) | 61.0 (2.65)
  CD4+ T cells, Day 8, 2 hours after EOI: number analyzed (Participants) | 26 | 57
  CD4+ T cells, Day 8, 2 hours after EOI | 103.4 (5.87) | 32.2 (2.52)
  CD8+ T cells, Day 1, 2 hours after EOI: number analyzed (Participants) | 20 | 57
  CD8+ T cells, Day 1, 2 hours after EOI | 95.2 (2.72) | 93.7 (3.06)
  CD8+ T cells, Day 4, 2 hours after EOI: number analyzed (Participants) | 23 | 54
  CD8+ T cells, Day 4, 2 hours after EOI | 111.1 (10.56) | 77.1 (4.33)
  CD8+ T cells, Day 8, pre-dose: number analyzed (Participants) | 26 | 54
  CD8+ T cells, Day 8, pre-dose | 101.8 (6.19) | 62.3 (2.68)
  CD8+ T cells, Day 8, 2 hours after EOI: number analyzed (Participants) | 26 | 57
  CD8+ T cells, Day 8, 2 hours after EOI | 103.0 (6.05) | 36.2 (2.52)

ADVERSE EVENTS:
Time Frame: Upto Month 24
Description: Safety was used for analysis which comprised of all participants who received any part of at least 1 infusion of study drug.
Arm/Group | Placebo | Otelixizumab
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/181
Serious Adverse Events (participants affected / at risk) | 6/91 | 15/181
Other Adverse Events (participants affected / at risk) | 81/91 | 173/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | Otelixizumab (N=181)
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Septic embolus (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 3
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | Otelixizumab (N=181)
Headache (Nervous system disorders) | 45 (117) | 155 (441)
Nausea (Gastrointestinal disorders) | 20 (32) | 60 (91)
Nasopharyngitis (Infections and infestations) | 29 (42) | 48 (83)
Fatigue (General disorders) | 20 (32) | 42 (58)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 (35) | 25 (35)
Vomiting (Gastrointestinal disorders) | 13 (15) | 35 (40)
Pyrexia (General disorders) | 10 (10) | 34 (45)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (27) | 21 (32)
Upper respiratory tract infection (Infections and infestations) | 10 (15) | 22 (29)
Lymphadenopathy (Blood and lymphatic system disorders) | 13 (20) | 18 (37)
Chills (General disorders) | 6 (9) | 24 (32)
Dizziness (Nervous system disorders) | 12 (20) | 18 (23)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (16) | 22 (83)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 19 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 20 (23)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 13 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 13 (16)
Sinusitis (Infections and infestations) | 4 (4) | 12 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 8 (13)
Blood creatine phosphokinase increased (Investigations) | 6 (6) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (11)
Pharyngitis (Infections and infestations) | 9 (13) | 4 (4)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (17)
Malaise (General disorders) | 2 (2) | 10 (13)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (15)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (11)
Insomnia (Psychiatric disorders) | 5 (5) | 5 (6)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (7)
Viral infection (Infections and infestations) | 6 (9) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.